CLINICAL TRIAL: NCT05933590
Title: Cervical Joint Repositioning Error in Different Head Positions Among Individuals With Chronic Migraine: A Cross-Sectional Study
Brief Title: Cervical Repositioning Error in Chronic Migraine
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/2820236
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Migraine; Chronic Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Migraine Group: This group consists of 25 individuals diagnosed with chronic migraine. They will undergo cervical joint repositioning error assessment in different head positions.
  Interventions: Diagnostic Test: Cervical Joint Repositioning Error Assessment
- Control Group: This group consists of 25 age-matched healthy controls without a history of migraine. They will undergo the same cervical joint repositioning error assessment in different head positions.
  Interventions: Diagnostic Test: Cervical Joint Repositioning Error Assessment

INTERVENTIONS:
Diagnostic Test: Cervical Joint Repositioning Error Assessment — The cervical joint repositioning error assessment is a non-invasive diagnostic test used to measure the ability of an individual to accurately reproduce a specific head position in different orientations (flexion, neutral position, 50% range of motion of left rotation, and 50% range of motion of right rotation). Participants in both the chronic migraine group and the control group will undergo this assessment using a digital inclinometer. The primary outcome of this study is the difference between the initial and repositioned cervical joint angles, measured in degrees.

SUMMARY:
This study examines cervical joint position sense in individuals with chronic migraine vs. healthy controls. The ability to reposition the cervical spine after active movement will be evaluated in different head positions. Impaired proprioception and motor control is hypothesized in the migraine group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 years old
* Diagnosis of chronic migraine (for the chronic migraine group)
* No history of migraine (for the control group)

Exclusion Criteria:

* History of cervical spine pathology
* Neurological deficits unrelated to migraine
* Current pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals aged 18-65 years old, with and without chronic migraine.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Cervical Joint Repositioning Error Assessment | Baseline
  The cervical joint repositioning error assessment is a non-invasive diagnostic test used to measure the ability of an individual to accurately reproduce a specific head position in different orientations (flexion, neutral position, 50% range of motion of left rotation, and 50% range of motion of right rotation). Participants in both the chronic migraine group and the control group will undergo this assessment using a digital inclinometer.The primary outcome of this study is the difference between the initial and repositioned cervical joint angles, measured in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No